CLINICAL TRIAL: NCT04233476
Title: Safety and Efficacy of 99mTc-hydrazinonicotinamide-PEG4-E[PEG4-c(RGDfk)]2 (99mTc-3PRGD2) SPECT/CT for Integrin αVβ3 Imaging of Lung Cancer and Mapping Lymph Node Metastases: A Prospective Multicenter, Self-controlled, Phase 3 Trial
Brief Title: 99mTc-3PRGD2 SPECT/CT for Integrin Imaging of Lung Cancer
Acronym: TRIIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RDO Pharm. (Industry)
Collaborators: Beijing Pharbers Genesis Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FSRDA201901
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Lung Cancer; Lymph Node Metastasis
Keywords: 99mTc-3PRGD2; Integrin ανβ3; lung cancer; lymph node metastasis
MeSH Terms: conditions — Lung Neoplasms; Lymphatic Metastasis | interventions — Technetium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 99mTc-3PRGD2 injection for SPECT/CT imaging, with 18F-FDG PET/CT for head-to-head comparison. (Experimental): Participants will receive a single-dose intravenous injection of 99mTc-3PRGD2 at a dosage of approximate 11.10 MBq (0.30 mCi) per kilogram body weight. Whole-body planar scan and chest SPECT/CT imaging will be performed 40-50 min later. Chest low-dose spiral CT (120 kV, 50 mAs) will be used for attenuation correction and anatomical localization.
  The conventional metabolic imaging by 18F-FDG PET/CT of the same patients within one week will be used for a self-controlled head-to-head comparison.
  Interventions: Drug: 99mTc-3PRGD2 injection

INTERVENTIONS:
Drug: 99mTc-3PRGD2 injection — A diagnostic drug targeting integrin αvβ3, technetium-99m [99mTc] labeled hydrazinonicotinamide-PEG4-E[PEG4-c(RGDfk)]2 (99mTc-3PRGD2), will be intravenously injected to the participants for imaging of lung cancer and mapping lymph node metastasis via single photon emission computed tomography/ X-ray computed tomography (SPECT/CT) .
  Other Names: Technetium-99m [99mTc] labeled hydrazinonicotinamide-PEG4-E[PEG4-c(RGDfk)]2

SUMMARY:
This is a prospective, multicenter, self-controlled phase 3 clinical trial designed to evaluate the safety and efficacy of an integrin αVβ3-targeted imaging, 99mTc-3PRGD2 SPECT/CT, for diagnosis of lung cancer and mapping the lymph node metastases. The pathological results will be considered as the gold standard and the conventional metabolic imaging by 18F-FDG PET/CT will be used for a head-to-head comparison. The primary objective of this study is to evaluate the efficacy of 99mTc-3PRGD2 SPECT/CT in mapping of lymph node metastasis according to the nodal mapping system released by the International Association for the Study of Lung Cancer in 2009 (IASLC-2009). The secondary objectives include evaluation of 99mTc-3PRGD2 SPECT/CT in detection of lung cancer and the safety of 99mTc-3PRGD2 injection in human beings.

DETAILED DESCRIPTION:
Accurate evaluation of lymph node metastasis plays a pivotal role in optimizing the surgical intervention and other precision treatments for lung cancer. CT-based nodal staging of lung cancer has limitation due to its low sensitivity, which relies on variations in tumor's size and structure. 18F-FDG PET/CT demonstrates low specificity owing to the nonspecific uptake in inflammatory lymph nodes, typically necessitating additional invasive mediastinal staging. Integrin αVβ3-targeted imaging could potentially bridge this existing technical gap. As a member of integrin family, integrin αVβ3 plays a crucial role in mediating tumor formation, invasion, metastasis, and angiogenesis. Therefore, integrin αVβ3 is an attractive target for tumor diagnosis and therapy. However, as of today, no drug has been approved for either diagnosis or therapy by targeting integrin αVβ3.

A diagnostic drug targeting integrin αvβ3, technetium-99m [99mTc] labeled hydrazinonicotinamide-PEG4-E[PEG4-c(RGDfk)]2 (99mTc-3PRGD2), has been developed for imaging of lung cancer and other tumors via single photon emission computed tomography/ X-ray computed tomography (SPECT/CT). After intravenous injection into the body, 99mTc-3PRGD2 is expected to be specifically taken up by integrin αVβ3-positive tumors. The images obtained by SPECT/CT will be used for diagnosis and evaluation of the tumors, thereby guiding the individualized treatments including surgical intervention.

A prospective, multicenter, self-controlled phase 3 clinical trial is designed to evaluate the safety and efficacy of an integrin αVβ3-targeted imaging, 99mTc-3PRGD2 SPECT/CT, for diagnosis of lung cancer, with mapping the lymph node metastases as the primary objective. The secondary objectives include evaluation of 99mTc-3PRGD2 SPECT/CT in detection of lung cancer and the safety of 99mTc-3PRGD2 injection in human beings. The pathological results will be considered as the gold standard and the conventional metabolic imaging by 18F-FDG PET/CT will be used for a head-to-head comparison.

More than 400 patients with suspected lung cancer are designed to be recruited from 11 medical centers. Participants who meet the inclusion and exclusion criteria will be recruited to undergo SPECT/CT planar scan and chest tomography after intravenous injection of 99mTc-3PRGD2 at a dose of 0.3 mCi/kg. They will also undergo 18F-FDG PET/CT within a week. Among them, the patients who successfully complete safety tests are included into the safety analysis set.

At least 270 participants are expected to undergo lung lobectomy and lymph node station resection within 2 weeks after the 99mTc-3PRGD2 SPECT/CT. Their pathological results will be collected and used as the gold standard to evaluate the diagnostic efficacy of 99mTc-3PRGD2 SPECT/CT for diagnosis of lung tumors and lymph node metastases, with a head-to-head comparison with 18F-FDG PET/CT. Those patients who undergo lung surgery and lymph node resection within two weeks after the 99mTc-3PRGD2 SPECT/CT will be included into the efficacy analysis set to evaluate the efficacy of the imaging method in diagnosis of lung cancer and mapping the lymph node metastases.

ELIGIBILITY:
Inclusion criteria

Participants must meet all of the following inclusion criteria to be eligible for this study:

1. Voluntarily participate and sign the Informed Consent Form;
2. Age ≥18 years old;
3. Diagnostic CT shows that the longest diameter of the tumor occupying the lung is ≥1.5 cm and the shortest diameter is ≥1.0 cm;
4. 18F-FDG PET/CT examination shows tumor occupancy in the lungs, with positive hilar and/or mediastinal lymph nodes on either enhanced CT or 18F-FDG PET/CT;
5. Willing and be able to follow scheduled visits, treatment plans, and laboratory tests;
6. Clinical laboratory examination and other indicators are within the normal range or abnormal but do not affect related examinations and treatments.

Exclusion criteria

Patients who have any of the following are not eligible for enrollment:

1. Female patients who plan of pregnant within 6 months, or in pregnant or lactating;
2. Allergic to the test drugs, have allergic constitution, or are allergic to multiple drugs;
3. Contrast-enhanced CT examination shows ground-glass nodules without solid components;
4. Before injecting 18F-FDG, the fasting blood glucose level exceeds 7.0 mmol/L (tested by rapid blood glucose meter);
5. Body weight exceeds 100 kg;
6. With claustrophobia;
7. Cannot tolerate raising their arms and lying on the scanner bed for 15-30 min;
8. Those the investigator believes not suitable to participate in this clinical trial;
9. Those who are currently participating in another clinical trial or have participated in other clinical trials within the past 3 month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 409 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2021-05-08 (Actual)

PRIMARY OUTCOMES:
Evaluate whether the diagnostic specicity of 99mTc-3PRGD2 SPECT/CT is superior to that of 18F-FDG PET/CT in mapping lymph node metastasis of lung cancer in the same group of patients. | From the informed consent of the first participant to 2 weeks after the intervention of the last participants or until the last participant accepted surgery within 2 weeks
  Using the pathological results as the gold standard, calculate the specificity of 99mTc-3PRGD2 SPECT/CT in mapping of lymph node metastasis of lung cancer according to the nodal mapping system released by the International Association for the Study of Lung Cancer in 2009 (IASLC-2009), and compared it head-by-head with that of the conventional metabolic imaging by 18F-FDG PET/CT in the same group of patients. And then assess if the specificity of 99mTc-3PRGD2 SPECT/CT is superior to that of 18F-FDG PET/CT.

SECONDARY OUTCOMES:
Diagnostic accuracy, sensitivity, positive predictive value and negative predicive value of 99mTc-3PRGD2 SPECT/CT in mapping lymph node metastasis of lung cancer, with a head-to-head comparison to 18F-FDG PET/CT. | From the informed consent of the first participant to 2 weeks after the intervention of the last participants or until the last participant accepted surgery within 2 weeks
  Evaluate the diagnostic accuracy, sensitivity, positive predictive value and negative predicive value of 99mTc-3PRGD2 SPECT/CT in mapping of lymph node metastasis of lung cancer according to the nodal mapping system released by the IASLC-2009. The pathological results will be considered as the gold standard and the conventional metabolic imaging by 18F-FDG PET/CT will be used for a head-to-head comparison.
Efficacy of 99mTc-3PRGD2 SPECT/CT in diagnosis of lung cancer, with a head-to-head comparison to 18F-FDG PET/CT. | From the informed consent of the first participant to 2 weeks after the intervention of the last participants or until the last participant accepted surgery within 2 weeks
  With the pathological diagnoses as the gold standard, the diagnostic values of 99mTc 3PRGD2 SPECT/CT will be obtained and the conventional metabolic imaging by 18F-FDG PET/CT will be used for a head-to-head comparison.
Incidence of adverse events for safety evaluation of 99mTc-3PRGD2 injection and SPECT/CT imaging in human beings | From the informed consent of the first participant to 2 weeks after the intervention of the last participants or until the last participant accepted surgery within 2 weeks
  Number of participants with adverse events, including treatment-emergent abnormality in vital sign measurements, physical examinations, 12-lead electrocardiogram report, or clinical laboratory tests (routine blood tests, blood biochemical tests, routine urine tests, etc). The relevant adverse reactions emerged during the study will be questioned or examined, and then recorded in detail to evaluate the safety of 99mTc-3PRGD2 SPECT/CT in the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (11):
- China (11):
  - Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shengyang, Liaoning
  - Renji Hospital of Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - First Hospital of Shanxi Medical Universit, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No
Shared according to requests and permission.